CLINICAL TRIAL: NCT06166628
Title: Efficacy of Genicular Artery Embolization Compared to Sensory Deinnervation for the Treatment of Symptomatic Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Genicular Artery Embolization vs Nerve Ablation Intervention (GENI) for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Clinkard (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor-Investigator, David Clinkard, Anesthesiologist, Department of Anesthesiology and Perioperative Medicine, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6038931
Record Dates: First submitted 2023-11-21; First posted 2023-12-12 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis
Keywords: Artery embolization; Nerve ablation; Genicular Artery Embolization
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Genicular artery embolization (Active Comparator): Genicular artery embolization will be performed by board certified Interventional Radiologists in the interventional radiology angiography suite at Kingston General Hospital. Patients will be blinded to which procedure they have been randomized too, careful language will be used by the clinical and research team throughout the procedure to not compromise the blinding. Patients will be positioned supine on the procedure table. The affected knee will be prepped and draped using standard sterile technique and 1-2cc of 1% lidocaine will be administered to the area for local anesthetic. A drape will be placed such that the patient is unable to see the affected knee during the procedure. Geniculate artery embolization will be performed via an intraarterial access and use of embolization microspheres injected into the hypervascular arteries feeding the knee joint.
  Interventions: Procedure: Geniculate artery embolization
- Genicular nerve phenol nerve ablation (Active Comparator): Genicular nerve phenol nerve ablation All procedures will be performed by a fellowship trained interventional pain physician in a fluoroscopy suite in Hotel Dieu Hospital using sterile precautions. Patients will be blinded to which procedure they have been randomized too, careful language will be used by the clinical and research team throughout the procedure to not compromise the blinding. IV access and saline lock obtained per our usual clinic protocol. Patients will be positioned supine on the procedure table. The affected knee will be prepped and draped using standard sterile technique and 1-2cc of 1% lidocaine will be administered to the area for local anesthetic. Phenol nerve ablation will be performed via ultrasound guidance.
  Interventions: Procedure: Genicular nerve phenol nerve ablation
- Sham procedure (Sham Comparator): The sham procedure will be performed by a fellowship trained interventional pain physician in a fluoroscopy suite in Hotel Dieu Hospital using sterile precautions. Patients will be blinded to which procedure they have been randomized too, careful language will be used by the clinical and research team throughout the procedure to not compromise the blinding. IV access and saline lock obtained per our usual clinic protocol. The patient will be placed supine, and the appropriate knee prepped and draped using appropriate sterile technique . A drape will be placed such that the patient is unable to see the affected knee during the procedure.
  Interventions: Procedure: Skin infiltration of 2cc of 0.25% bupivacaine at the knee

INTERVENTIONS:
Procedure: Geniculate artery embolization — Femoral arterial access will be obtained under ultrasound guidance. An angiographic catheter will then be advanced to the distal superficial femoral artery. Angiography will be performed to identify the appropriate genicular branches supplying the regions of hyperemia. A microcatheter (1.7-2.4-French) will then be advanced super-selectively into the genicular arteries and 100-300 um EmboSpheres (Merit Medical) will be injected under fluoroscopic guidance. Multiple geniculate arteries may be embolized until neovascularity is no longer seen and pathologic hyperemia is resolved. A repeat lower extremity angiogram will be performed to evaluate for success of embolization and to exclude complication. The catheter and sheath will then be removed, and hemostasis will be achieved using an AngioSeal (Terumo Vascular Interventions) vascular closure device.
  Arms: Genicular artery embolization
Procedure: Genicular nerve phenol nerve ablation — A high frequency ultrasound probe and anatomic landmarks will be used to identify the location of the genicular nerves as well as the nerves to the vastus lateralis, vastus intermedius and vastus medialis. Utilizing an in or out of plane approach as necessary, a 25 g spinal needle will be advanced to the appropriate location after skin anesthesia with 1cc of 1% lidocaine. After negative aspiration, 2 cc of 6% phenol will be injected at each location with an end target of fascial expansion under the relevant fascial plane.
  Arms: Genicular nerve phenol nerve ablation
Procedure: Skin infiltration of 2cc of 0.25% bupivacaine at the knee — A high frequency ultrasound probe and anatomic landmarks will be used to identify the location of the genicular nerves as well as the nerves to the vastus lateralis, vastus intermedius and vastus medialis will be identified. Utilizing an in or out of plane approach as necessary, a 25 g spinal needle will be advanced to the appropriate location after skin anesthesia with 1cc of 1% lidocaine. After negative aspiration, 1.5 cc of sterile saline will then be injected at each location.
  Arms: Sham procedure

SUMMARY:
The genicular artery embolization vs nerve ablation intervention (GENI) knee OA study is a three-arm randomized controlled trial to evaluate symptoms of knee osteoarthritis (OA) in patients after receiving one of three interventions: sham procedure, geniculate artery embolization (GAE) or genicular nerve phenol nerve ablation (PNA).

The main question[s] the study aims to answer are:

* Does GAE or genicular nerve PNA result in OA symptom alleviation compared to sham procedure?
* Are there molecular or imaging biomarkers that aid in predicting treatment response for GAE or genicular nerve PNA?

Subjects (N=150) patients with knee OA, resistant to non-surgical treatment for at least 3 months will be randomized 1:1:1 to either after GAE, genicular nerve PNA or sham procedure. Clinical outcomes will be measured using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and 11-point numerical rating scale (NRS) for pain completed at baseline, 1 month, 3 months, and 6 months and then every 6 months for either two years or until the time of total knee arthroplasty (TKA) surgery.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is a common and debilitating disease. Advanced disease can be treated with total knee arthroplasty (TKA), however knee OA that is either resistant to non-surgical options, or where surgical options are not available, represents a specific management challenge. Genicular artery embolization (GAE) and genicular nerve phenol nerve ablation (PNA) have emerged as potentially successful treatments to reduce knee OA symptoms, however, to date no randomized controlled trials have been completed comparing the two procedures.

The purpose of this study is to compare the clinical outcomes of GAE to genicular nerve PNA for chronic knee pain in patients with knee OA. Further, molecular biomarkers and imaging will be taken pre- and post-procedure to evaluate if immune-mediated neuroinflammation and angiogenesis can be helpful in predicting treatment response.

This single center randomized controlled trial will be conducted to determine if GAE, genicular nerve PNA, or sham procedure is associated with a clinically significant alleviation of knee OA symptoms. The investigators aim to include 150 participants in this study over the course of 24 months randomized 1:1:1 to receive either GAE, genicular nerve PNA, or sham procedure.

After eligibility is confirmed and consent is obtained, a baseline assessment will be conducted including baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and 11-point numerical rating scale (NRS) for pain scores. Participants will receive a knee 3T MRI with gadolinium contrast and 0.5 - 5 mL of synovial fluid will be aspirated for baseline analysis. Participants will receive Fitbit motion trackers to quantify activity levels throughout the study.

Study procedures will be performed by either a qualified Interventional Radiologist or fellowship-trained Anesthesiologist, depending on which study arm subjects randomized to.

Approximately 3 months after the procedure, repeat WOMAC and NRS scores will be obtained, in addition to repeat 3T MRI with gadolinium contrast and knee aspirate of 0.5 - 5 mL of synovial fluid. Additional questions pertaining to knee-specific analgesia use, adverse events from the procedure, or any concerns will be addressed and noted at this time.

Participants will be followed up by phone by a blinded member of the research team 6 months after the procedure and every 6 months thereafter for 2 years or until the time of TKA surgery (if applicable). During phone calls, questions relating to knee-specific analgesia use will be asked and repeat WOMAC and NRS scores will be acquired.

Data for this study includes: demographic information, knee-specific analgesia use, which procedure was performed, knee 3T MRI with gadolinium contrast, WOMAC scores, NRS pain scores, knee synovial fluid cytokine/chemokine biomarker analysis, and procedure-specific adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years
* Able to provide informed consent
* Knee pain due to osteoarthritis for at least 6 months
* Pain refractory to conservative therapies (oral medication, or physical therapy, or activity modification) for at least 3 months with a desire for TKA
* Candidate for TKA at Hotel Dieu Hospital Site
* Able to comply with all treatments and protocol follow-up visits

Exclusion Criteria:

* Current local infection
* Systemic or joint centered inflammatory disease (ie rheumatoid arthritis, Lupus, multiple sclerosis or other autoimmune diseases)
* Current use of systemic immunosuppression therapy
* Known lower extremity vascular disease or lower extremity symptoms thought to be secondary to arterial vascular disease (eg claudication, ischemic rest pain)
* Irreversible coagulopathy
* Renal dysfunction as defined by GFR (eGFR) of <30 obtained within the past 60 days
* Contraindication for MR Imaging (such as claustrophobia, metallic fragment or foreign bones, implants or prosthesis)
* IV CT and/or MRI contrast allergy characterized by anaphylaxis or anaphylactoid reactions
* Pregnancy or women of childbearing potential not currently on a medically acceptable method of birth control

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in knee pain/functionality post geniculate artery embolization versus nerve ablation vs sham | 3 months
  Overall efficacy of treatment as determined by a clinically significant reduction in Western Ontario and McMaster University Osteoarthritis Index (WOMAC) questionnaire of 20 points or more.
  The WOMAC is a questionnaire evaluating knee osteoarthritis with subcategory scores for pain (0-20 points), stiffness (0 - points), physical function (0-8 points), and sum total score (0-96 points) with higher values indicating more severe symptoms.

SECONDARY OUTCOMES:
Changes in numerical rating scale pain scores post geniculate artery embolization versus nerve ablation vs sham | 3 and 6 months
  Assessment of changes in the 11-point numerical rating scale (NRS) for pain where 0 indicates no pain and 10 indicates maximal pain. A decrease of 2 points or more from baseline will be considered a minimal clinically important decrease.
Assessment of desire for total knee arthroplasty post geniculate artery embolization versus nerve ablation vs sham | 3 and 6 months
  Participants will be asked whether they feel their current symptoms are still sufficiently severe that they would like to proceed with knee replacement.
Evaluation of MRI | 3 months
  Assessment of change in MRI features using whole-organ magnetic resonance imaging score (WORMS) of the knee in osteoarthritis.
  The WORMS assesses 14 subregions of the knee divided by anatomical landmarks. In each subreagion, 14 types of structural changes are assessed. This include: cartilage integrity, subarticular bone marrow edema, subarticular cysts, subarticular bone flattening, marginal ostophytes, medial-lateral meniscal tears, integrity of the anterior and posterior cruciate ligaments, integrity of the medial and lateral collateral ligaments, synovitis/effusion, loose body, and periarticular cysts/bursitis.
  The sum of all anatomic regions and structural feature scores is the total WORMS score from 0 - 332 with a higher score indicating MRI features associated with more severe osteoarthritis.
Evaluation of Synovial Fluid | 3 months
  Synovial fluid samples taken before study intervention and 3 months post intervention will be compared.
  Protein from each sample will be assessed using multiplex Luminex analysis for targeted inflammatory protein expression using EMD Millipore Human Cytokine/Chemokine/Growth Factor panel.

CONTACTS AND LOCATIONS:
Overall Officials: David Clinkard, MD, Principal Investigator — Queen's University; Alexandre Menard, MD, Principal Investigator — Queen's University; Steve Mann, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No